CLINICAL TRIAL: NCT00895479
Title: A Phase III, Randomized, Controlled, Open Label, Multicenter Study of the Efficacy and Safety of Trinam® (EG004); an Assessment of Primary Unassisted Patency and Survival of Vascular Access Grafts in Hemodialysis Patients With End Stage Renal Disease
Brief Title: Adenovirus Vascular Endothelial Growth Factor (VEGF) Therapy in Vascular Access - Novel Trinam AGainst Control Evidence
Acronym: AdV-VANTAGE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic reasons. Seeking partner for future development.
Sponsor: Ark Therapeutics Ltd (Industry)
Responsible Party: Director of Research and Development, Ark Therapetics Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ark 103
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease; ESRD; Hemodialysis; Access Graft
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trinam (Experimental): Graft placement plus Trinam therapy
  Interventions: Procedure: Graft placement surgery plus Trinam therapy
- Control (No Intervention): Graft placement surgery alone

INTERVENTIONS:
Procedure: Graft placement surgery plus Trinam therapy — Trinam arm: graft placement surgery plus 1ml perivascular administration of Trinam vector.
  Control arm: graft placement surgery
  Arms: Trinam

SUMMARY:
Patients in renal failure on hemodialysis depend on adequate and sustained vascular access. This can be achieved by surgical placement of a synthetic polytetrafluoroethylene (PTFE) graft. These patients frequently experience graft complications arising from the development of smooth muscle cell (SMC) neointimal hyperplasia in the proximity of the graft-vein anastomosis. Such complications eventually lead to stenosis, access thrombosis and graft failure. Trinam® is being developed to prolong graft survival. It is a combination product consisting of a replication deficient Adenovirus containing the human Vascular Endothelial Growth Factor D (Ad-VEGF-D) gene and a biodegradable local delivery device (collar) made of collagen. At the end of the surgical procedure to insert the PTFE graft the collagen collar is applied around the anastomosis and sealed with a collagen surgical sealant. This procedure creates a reservoir between the site of anastomosis and the collagen collar. The adenoviral vector is then injected into this reservoir, localizing the expression of the transgene to the site of the anastomosis. Expression of VEGF-D has been shown to have a vascular protective role and inhibit SMC neointimal proliferation, therefore expression of VEGF-D should prolong graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease undergoing either initial placement or replacement (after failure of previous vascular access) of an end-to-side or end-to-end 6.0 mm synthetic PTFE arteriovenous hemodialysis access arm graft.
* Male or female aged 18 years or over.
* Patients who signed the informed consent form.
* Patients who are expected to undergo dialysis at nominated facilities for the duration of the study.
* Patients who have agreed to participate in the additional four year gene therapy safety monitoring.
* Patients who are willing to agree they will not have a kidney transplant for four weeks post treatment with Trinam®.
* Patients who have undergone arterial and venous mapping to ensure an adequate and appropriate access site is available for placement of either an end-to-side or an end-to-end 6.0 mm synthetic PTFE arteriovenous hemodialysis access arm graft with or without the addition of Trinam®.

Exclusion Criteria:

* Patients who are unable to understand and sign the consent form.
* Patients undergoing surgical revision of an existing graft.
* Exclude patients from the study if they have moderate or severe macular edema moderate or severe proliferative diabetic retinopathy
* Current diagnosis of cancer with exception of non-melanoma skin cancers.
* Hepatic dysfunction defined as AST and / or ALT > 2 times the Upper Limit of Normal.
* Diabetic patients with Hemoglobin A1C value of >10%.
* White blood cell (WBC) count < 2.0 x 109/L.
* Prior anticoagulant therapy within 14 days prior to surgery is an exclusion.
* Known sensitivity to collagen.
* Pregnancy, lactation or lack of effective contraception both in women and in men of childbearing potential.
* Previous participation in any Trinam® study.
* Receipt of any investigational drug within 30 days prior to study enrollment or participation in any concurrently running trial involving investigational intervention.
* Any medical or psychiatric condition that compromises the ability to participate in the study.
* Known or suspected drug or alcohol abuse in the past six months.
* Life expectancy of less than one year.
* Known immunodeficiency disease.
* Known chronic hepatitis of viral or non-viral etiology and / or a history of decompensated liver failure of any etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Primary Unassisted Patency | 18 Months

SECONDARY OUTCOMES:
Graft Survival. Number and rate of graft interventions. | 2.5 years

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Long Beach VA Healthcare System, Long Beach, California
  - Four Rivers Clinical Research Inc, Paducah, Kentucky
  - Baton Rouge General Hospital, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - St Luke's Roosevelt Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Division of Nephrology, Columbus, Ohio
  - Texas Tech University Medical Center, Lubbock, Texas
  - Harborview Medical Center, Seattle, Washington